CLINICAL TRIAL: NCT04771910
Title: Study of the Skin Microbiome and the Potential of a Topical Probiotic Cream for Atopic Dermatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Collaborators: YUN NV (Industry)
Responsible Party: Principal Investigator, ethisch.comite@uza.be, Prof. Dr. Sarah Lebeer, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B3002020000099
Record Dates: First submitted 2020-08-14; First posted 2021-02-25 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Atopic Dermatitis
Keywords: Skin microbiome; Probiotics; Lactobacillus spp.
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: All AD patients will receive both treatments (verum and placebo). Verum cream will be applied on one side of the body (elbow or knee cavities), the placebo cream on the other side.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical cream with live probiotic bacteria (YUN) (Experimental): Patients with atopic dermatitis using topical cream with live probiotic bacteria
  Interventions: Other: Topical cream with live probiotic bacteria
- Placebo cream (YUN) (Placebo Comparator): Patients with atopic dermatitis using placebo cream (same formulation as probiotic cream except live probiotic bacteria)
  Interventions: Other: Placebo cream

INTERVENTIONS:
Other: Topical cream with live probiotic bacteria — Application of the probiotic cream once a day, for approximately 8 weeks on one side of the body (elbow or knee cavity; decided by doctor in advance, same as placebo cream). Assessment before product use (T0), after 4 and 8 weeks of product use (T4w and T8w, respectively) and after 4 weeks without product use (T12w).
  Other Names: ACN cream (YUN)
  Arms: Topical cream with live probiotic bacteria (YUN)
Other: Placebo cream — Application of the placebo cream (same formulation as probiotic cream except live probiotic bacteria) once a day, for approximately 8 weeks on one side of the body (elbow or knee cavity; decided by doctor in advance, same as probiotic cream). Assessment before product use (T0), after 4 and 8 weeks of product use (T4w and T8w, respectively) and after 4 weeks without product use (T12w).
  Arms: Placebo cream (YUN)

SUMMARY:
The skin microbiome of atopic dermatitis patients and healthy volunteers will be studies by collecting and analysing skin swabs on different timepoint. Additional, effort will be made to isolate and characterize Lactobacillus spp. and other beneficial micro-organisms on the skin. Second aim of this study is to evaluate a topical probiotic cream in atopic dermatitis treatment. A double-blind placebo-controlled intervention study will be performed in parallel with the skin microbiome analysis. Both clinical effect on the symptoms of atopic dermatitis and effect on the skin microbiome and survival of beneficial bacteria on the skin will be evaluated.

DETAILED DESCRIPTION:
Probiotics are live micro-organisms which when administered in adequate amounts can exert a health benefit on the host. This health-promoting effects have been extensively studied in the gastrointestinal niche but it becomes more and more clear that other niches are also interesting for the potential of probiotics. Recent breakthroughs in 'next generation sequencing' (NGS) technologies are making it now possible to map the microbiota after DNA extraction, which is very interesting for bacteria that are not or difficult to cultivate. The research into the microbiota of the skin with such new NGS technologies shows that there is also an equilibrium in the skin composition of the microbiota and that there is a disturbance of the skin microbiota in atopic dermatitis (AD). The etiology of AD is complex, with the manifestation of the disease being influenced by various genetic and immune mechanisms acting in concert with environmental factors. A reduction in the skin microbial diversity is often observed and flares are characterized by an abundance of skin pathobionts such as Staphylococcus aureus. Therefore, topical probiotic strains could have a positive effect on the skin microbiome and function by inhibiting pathogens, restoring the skin microbiome and/or barrier function and executing anti-inflammatory effects on the skin cells. The main objectives of this study are to analyse the skin microbiome in healthy volunteers and patients AD to obtain in depth data of the composition of the skin microbiome and identify possible biomarkers for AD. In parallel, a double-blind placebo-controlled study with topically applied live lactobacilli will be performed to give more insights in the working mechanisms of lactobacilli on AD skin. More specifically to evaluate the effect of the 'live' Lactobacillus species as 'active ingredient' in relation to acne symptoms and skin microbiome modulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atopic dermatitis and healthy volunteers

Exclusion Criteria AD patients:

* no use of topical antibiotics and/or corticosteroids within 2 weeks before the start
* no use of oral antibiotics within 1 month before the start
* no immunodeficiency disease

Exclusion Criteria Healthy Population:

* no use of topical antibiotics and/or corticosteroids within 2 weeks before the start
* no use of oral antibiotics within 1 month before the start
* no immunodeficiency disease
* no history of atopic dermatitis or other inflammatory skin disorders

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in skin microbiome composition | AD patients: skin swabs at baseline,4 and 8 weeks of product use and 4 weeks without product use (total 12 weeks). Healthy volunteers: skin swab at baseline and after 12 weeks (no product use)..
  Extraction of microbial DNA out of skin swabs. Analysis of differences in bacterial communities colonizing the skin between healthy individuals and AD patients measured via Next Generation Sequencing techniques and qPCR assays.
Change from baseline in AD severity scoring based on Eczema Area and Severity Index | AD patients: skin swabs at baseline,4 and 8 weeks of product use and 4 weeks without product use (total 12 weeks). Healthy volunteers: NA
  Evaluation of atopic dermatitis symptoms via a scoring system based on Eczema Area and Severity Index (EASI). The EASI will be adjusted to the limited area of elbow or knee cavities.
Change from baseline in itching via Visual Analogue Scale | AD patients: skin swabs at baseline,4 and 8 weeks of product use and 4 weeks without product use (total 12 weeks).
  The effect of the treatment of itching of the skin caused by atopic dermatitis lesions will be evaluated using Visual Analogue Scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Lebeer, Prof, Principal Investigator — Universiteit Antwerpen; Margo Hagendorens, Prof, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No